CLINICAL TRIAL: NCT06326905
Title: Addressing Inactive Kidney Transplant Waitlist Status Through Adapting a Tailored Psycho-Social-Environmental Program
Brief Title: CAPABLE Transplant
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00437750; K23DK133677-01A1 (NIH)
Record Dates: First submitted 2024-03-18; First posted 2024-03-22 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Quality of Life; Depression; End Stage Renal Disease; Disability Physical
Keywords: Activities of Daily Living; Instrumental Activities of Daily Living; Physical Function; Executive Function; Home; Intervention; Kidney Transplant; End Stage Renal Disease
MeSH Terms: conditions — Depression; Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Waitlist Control Trial
Who Masked: Outcomes Assessor
Masking Description: The assessment collector will be blinded as to whether a participant is in the intervention or waitlist group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Open Label Pilot (Experimental): The Open Label Pilot will include testing the CAPABLE Transplant intervention with 3 individuals on the waitlist.
  Interventions: Behavioral: CAPABLE Transplant- Open Label Pilot
- Randomized Control Pilot- Intervention Arm (Experimental): After the open label pilot, 20 participants will be randomized to the CAPABLE Transplant intervention. They will be assessed at baseline, after the 4 month intervention, and after the waitlist control arm.
  Interventions: Behavioral: CAPABLE Transplant- Randomized Control Trial
- Randomized Control Pilot- Waitlist Control Arm (Active Comparator): The waitlist control group, 20 participants, will receive the intervention after they have served as controls to the immediate treatment group, ensuring all participants have access to the intervention.
  Interventions: Behavioral: CAPABLE Transplant- Randomized Control Trial

INTERVENTIONS:
Behavioral: CAPABLE Transplant- Open Label Pilot — As in CAPABLE, the delivery characteristics of CAPABLE Transplant consist of an assessment-driven, individually tailored package of interventions delivered over the course of 4 months by an occupational therapist (OT) (~6 home visits for ≤ 1hour), a registered nurse (RN) (~4 home visits for ≤ 1hour) and a handy worker (HW).
  Adaptations targeting those currently KT inactive will be made on a per-client basis as part of the open-label pilot. We will further refine and develop the intervention by receiving feedback from the open label pilot participants and CAPABLE clinicians who implemented the pilot to gain their perspective of the acceptability and feasibility of implementing the CAPABLE-Transplant intervention. Based on this feedback, the study team will have developed an adapted iteration of the prototype.
  Arms: Open Label Pilot
Behavioral: CAPABLE Transplant- Randomized Control Trial — As in CAPABLE, the delivery characteristics of CAPABLE Transplant consist of an assessment-driven, individually tailored package of interventions delivered over the course of 4 months by an occupational therapist (OT) (~6 home visits for ≤ 1hour), a registered nurse (RN) (~4 home visits for ≤ 1hour) and a handy worker (HW). Refinements based on the open label pilot results will be included.
  Arms: Randomized Control Pilot- Intervention Arm; Randomized Control Pilot- Waitlist Control Arm

SUMMARY:
The purpose of this mixed methods study is to adapt CAPABLE as CAPABLE Transplant to accomplish two things: 1) To resolve barriers to being classified as active on the Kidney Transplant (KT) waitlist, 2) as a surgical prehabilitation intervention targeting the pre-frail/ frail KT waitlist population. It consists of two phases- an open label pilot and a randomized waitlist control trial, and 3) pilot test the feasibility and acceptability for CAPABLE Transplant in symptom and waitlist specific metrics amongst low-income active kidney transplant waitlist candidates.

DETAILED DESCRIPTION:
CAPABLE is a multicomponent goal-directed program that reduces physical disability by working with the person and environment but has not been explored in prehabilitation research. The purpose of this study is to adapt CAPABLE, an existing evidence-based program for functionally and socio-economically vulnerable older adults, as a prehabilitation intervention for people with frailty awaiting KT.

As in CAPABLE, the delivery characteristics of CAPABLE Kidney Transplant consist of an assessment-driven, individually tailored package of interventions delivered over the course of 4 months by an occupational therapist (OT) (~6 home visits for ≤ 1hour), a registered nurse (RN) (~4 home visits for ≤ 1hour) and a handy worker (HW).

In earlier phases, research team members conducted preliminary activities to design the CAPABLE Kidney Transplant intervention using Human-Centered Design techniques.

This study will seek to accomplish two aims:

1. To iteratively refine the CAPABLE -Transplant prototype for those currently KT inactive or those who are active and low-income on the waitlist.
2. To pilot test the CAPABLE-Transplant intervention

The investigators will collect feedback during the open label pilot to further refine the intervention that will be tested as part of the randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

* Deceased Donor Waitlist
* ≥18 years old
* Community dwelling
* Current Inactive status or active and had been inactive in the last 18 months for cardiovascular disease, frailty, obesity, social support, mental health, incomplete testing OR Active on the waitlist and low-income

Exclusion Criteria:

* Living Donor Waitlist
* Severe cognitive impairment
* Inactivity expected to last > 3 months (eg cancer treatment)
* >4 hospitalizations in the last 12 months
* Current home nursing, physical or occupational therapy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2025-01-25 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Waitlist-status as assessed by data obtained by the National Kidney Registry | 0, 16 weeks, 32 weeks
  Death (any cause), Time Inactive
  Change of waitlist status (inactive to active, delisting)

SECONDARY OUTCOMES:
Change in self-efficacy as assessed by the Coping Self-Efficacy Instrument | Baseline, 16 weeks, 32 weeks
  Coping Self-Efficacy is a 13 item instrument on a scale of 0 ('can't do at all') to 10 ('certain can do'). A higher score indicates higher level of self-efficacy when implementing coping strategies. Score range 0-130.
Change in self-efficacy as assessed by the Self-Efficacy of Chronic Disease Management Instrument | Baseline, 16 weeks, 32 weeks
  Self-Efficacy of Chronic Disease Management Instrument is a 6 item instrument on a visual analog scale, ranging from 1 (not at all confident) to 10 (totally confident). Lower scores indicate lower self-efficacy as indicated by confidence. Score range 6-60.
Change in Pain as assessed by the Brief Pain Inventory | Baseline, 16 weeks, 32 weeks
  The Brief Pain Inventory - is a 4-item self-administered questionnaire used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning. The patient is asked to rate their worst, least, average, and current pain intensity, list current treatments and their perceived effectiveness, and rate the degree that pain interferes with general activity, mood, walking ability, normal work, relations with other persons, sleep, and enjoyment of life on a 10 point scale. For the 10 point scale, 0 indicated no pain and 10 indicates the worst imaginable pain. Score range 0-40.
Change in Depression as assessed by the Patient Health Questionnaire Depression Scale (PHQ-8) | Baseline, 16 weeks, 32 weeks
  The PHQ-8 contains 8 questions, with a 0-3 scale. A score of 10 or greater is considered major depression, 20 or more is severe major depression. Score range 0-30.
Change in Social engagement as assessed by the Lubben Social Network Scale | Baseline, 16 weeks, 32 weeks
  The Lubben Social Network Scale is a 7-item questionnaire that measures the size of social networks of family and friends. The score ranges between 0 and 30, with higher scores indicated more social engagement.
Change in Social engagement as assessed by the Krause-Borawski-Clark Support Interactions Scale | Baseline, 16 weeks, 32 weeks
  The Krause-Borawski-Clark Support Interactions Scale is a 10-item self-reported questionnaire that measures social interactions. The scale is broken down into different domains; scores range from very often (4); fairly often (3); once in a while (2); never (1) or binary-- satisfied (1) or not satisfied (0) depending on domain within the questionnaire. Items are summed to form a single composite score range 10-40, Higher scores on the scale is associated with better personal perception and social support.
Change in Fatigue/Quality of Life as assessed by the Kidney disease Quality of Life Scale | Baseline, 16 weeks, 32 weeks
  The Kidney disease Quality of Life Short Form is a 20-item self-report outcome measure for patients on dialysis. Higher scores indicate better health-related quality of life. Scores range from 0-100.
Change in Frailty as assessed by the Fried Frailty Phenotype | Baseline, 16 weeks, 32 weeks
  The Fried Frailty Phenotype contains 5 criteria: unintentional weight loss >10lbs >5% of body mass in the last year, weakness (handgrip strength measurement), exhaustion (based on the Center for Epidemiological Studies Depression Scale), slow gait (walking time over a distance), and low physical activity. People who had none of the criteria were considered non-frail, people who had 1 and 2 criteria were considered pre-frail, and people who had ≥3 criteria were considered frail.
Change in Health Team Communication as assessed by the CollaboRATE Scale Measure | Baseline, 16 weeks, 32 weeks
  The CollaboRATE scale measure is a 3 item self-report questionnaire on patient's shared decision making. It is scored on a 10-point anchored scale, ranging from 0 ("no effort was made") to 9 ("every effort was made"). Higher scores indicate more shared decision making.
Change in Function as assessed by Lawton & Brody's assessment of Instrumental Activities of Daily Living Scale | Baseline, 16 weeks, 32 weeks
  The assessment contains 8 questions with answers that are either a score of 0 or 1. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent) for women, and 0 through 5 for men to avoid potential gender bias.
Change in Function as assessed by the Katz Index of Independence in Activities of Daily Living | Baseline, 16 weeks, 32 weeks
  6 questions, each 1 point for a total score of 6. A score closer to 6 indicates high patient independence.

OTHER OUTCOMES:
Acceptability at endpoint of intervention assessed by survey | 16 weeks
  Score on Likert scale-based questions re: program content & structure satisfaction, willingness to recommend. Survey developed by study team.
Feasibility as assessed by qualitative questions | 16 weeks
  Open/ Close Ended Questions, Recruitment Rate, Completion Rate, Data Collection Rate, Mean time for survey administration, Withdrawal Rate, Cost. Questions developed by study team.
Fidelity as assessed by percent completion of intervention items | 16 weeks
  % tasks/ patient- directed content delivery per session for Nurse & Occupational Therapist, % completion of home modifications

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Hladek, PhD, Principal Investigator — Johns Hopkins School of Nursing
Locations (1):
- Johns Hopkins School of Nursing, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No